CLINICAL TRIAL: NCT06775340
Title: Study to Evaluate the Safety, Tolerability, Pharmacodynamics and Efficacy of RSS0343 Tablets in Patients With Non-cystic Fibrosis Bronchiectasis
Brief Title: Study of RSS0343 Tablets in Patients With Non-cystic Fibrosis Bronchiectasis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RSS0343-201
Record Dates: First submitted 2025-01-09; First posted 2025-01-15 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-01

CONDITIONS: Adolescent Asthma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RSS0343 Tabella (Experimental)
  Interventions: Drug: RSS0343 Tabella

INTERVENTIONS:
Drug: RSS0343 Tabella — RSS0343 tablets, oral;

SUMMARY:
Studies to evaluate the safety, tolerability, pharmacodynamics, and efficacy of RSS0343 tablets in patients with non-cystic fibrosis bronchiectasis

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old (including boundary values), male and female.
2. Female subjects weigh ≥45 kg and male subjects weigh ≥50 kg.
3. HRCT shows bronchiectasis affecting one or more lobes of the lung and is confirmed by the clinician as NCFB.
4. The expected survival is greater than 12 months.
5. Informed consent was signed before the trial.
6. Potentially fertile subjects voluntarily take appropriate contraceptive measures.

Exclusion Criteria:

1. Patients with pulmonary hypertension or chronic obstructive pulmonary disease (COPD) or asthma as determined by the investigators were the primary diagnosis were screened.
2. An active, symptomatic infection caused by respiratory viruses, including COVID-19, influenza viruses, etc.
3. Have psoriasis or lichen planus.
4. Have Wright's disease/keratosis or hemorrhagic keratosis, or reactive arthritis.
5. Have chlorine acne, large common warts, or keratodermatitis.
6. Has diabetic foot.
7. Have periodontal disease, oral infection, or loose teeth.
8. History of malignant tumor within 5 years prior to screening.
9. Screening subjects with a history of liver disease or currently receiving treatment for liver disease, including but not limited to acute or chronic hepatitis, cirrhosis, or liver failure.
10. Researchers consider any other unstable clinical disease.
11. Oral or inhaled antibiotics were received 4 weeks prior to first administration.
12. Immunosuppressants were administered 4 weeks before the first dose.
13. Received drugs within 4 weeks prior to screening that may cause hyperkeratosis of the skin.
14. Received live attenuated vaccine within 30 days prior to initial administration.
15. Participated in clinical trials of any medical device within 3 months prior to screening.
16. Active hepatitis B virus infection, active hepatitis C virus infection, or known HIV infection or known syphilis infection.
17. Drug abusers.
18. Current smoker or former smoker for less than 3 months.
19. Suspected allergy to the investigational product or any component of the investigational product, or severe allergy to any drug, food, toxin or other exposure.
20. Pregnant or lactating women.
21. The subjects were unable to complete the questionnaires due to their limited educational level, or neither the subjects themselves nor their families could fill in the subject log card.
22. The researchers determined that there were other circumstances that were not suitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The number of occurrences of AEs | Day 1 to Day56
the frequency of occurrence of AEs | Day 1 to Day56

SECONDARY OUTCOMES:
RSS0343 amount of tablets of their metabolites in the blood | Day7, Day14, Day21, Day 28
Changes in the concentrations of active neutrophil elastase (NE) in sputum | Day7, Day14, Day21, Day 28, Day 56
Changes in the concentrations of cathepsin G (CatG) in sputum | Day7, Day14, Day21, Day 28, Day 56
Changes in the concentrations of enzyme protease 3 (PR3) in sputum | Day7, Day14, Day21, Day 28, Day 56

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided